CLINICAL TRIAL: NCT04324957
Title: Scale Development ,Content Validation and Reliability Testing of Neonatal Cardio-pulmonary Outcome Measure (N-COM) in Neonates Admitted in Neonatal Intensive Care Unit
Brief Title: Neonatal Cardio-Pulmonary Outcome Measure
Acronym: N-COM
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/1524; U1111-1249-3550 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-06; First posted 2020-03-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Congenital Heart Defect; Respiratory Distress Syndrome in Premature Infant
Keywords: Heart defects; Pulmonary function test; Newborns
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neonatal cardio-pulmonary outcome measure used to assess cardio-pulmonary status — Neonatal cardio-pulmonary outcome measure will be used to assess overall status of pulmonaryand cardio-vascular system

SUMMARY:
Neonatal Cardio-Pulmonary outcome measure (N-COM) will be used to assess the overall status of pulmonary and cardiac vascular system of neonates in Neonatal Intensive Care Unit (NICU). There are many scales available which are helpful for assessing behavior, pain, and neurological status of neonates but there is no scale available till now which can help to assess cardio-pulmonary status of neonates.

DETAILED DESCRIPTION:
Background:

Neonatal Intensive care unit (NICU) is exclusively created to treat premature and fragile neonates. The neonates with intrauterine growth limitations with congenital heart defects and respiratory diseases are at increased risk of mortality. There are several scales to assess pain, behaviour, motor changes, growth and other components of neonates. In the past, no scale is available to evaluate the cardio-pulmonary status of the neonates in NICU.

Objectives:

The objective of the study is to develop an outcome measure for checking the cardio-pulmonary status of the neonate in the Neonatal Intensive care units (NICU), as Neonatal cardio-pulmonary outcome measure (N-COM) and to validate the domains of the scale, to check the reliability and minimum desirable change (MCID).

Methods:

This study includes mainly four stages. In the first stage, different domains will be developed for the scale (N-COM) and scale will be sent for content validation. The domains of the scale will be made through different scales and the items will be selected from previous scales and from interview with medical personal working in NICU.

The lacking domains in the previous scales will be noted. The items will be evaluated by expert panel, undergo revision and pilot testing will be done. On the basis of acceptance, the pilot testing will undergo for final revision. In the second stage, the content validation of the items will be done. The test re-test reliability and inter-rater reliability will be done in this stage. In the third stage, the standard error of measurement (SEM) will be determined and minimal detectable change (MCID) at 95% Confidence Interval (CI) will be established for the scale.

Data analysis:

The content validity will be estimated by Item-content validity index (I-CVI) and scale-content validity index (S-CVI). The items and domains in the N-COM scale will undergo intra-rater and test-retest reliability testing by intra-class correlation coefficient (ICC) and criterion-related validity by Spearman Rank correlation coefficient.

Discussion:

The Neonatal cardio-pulmonary outcome measure (N-COM) will be the first scale which will help to assess respiratory and cardiac problems in the neonates. This scale N-COM will provide the general status of the cardio-pulmonary system of neonates. This scale will help to document the pre -intervention and post-intervention changes in the cardio-pulmonary system of neonates. As the item and domain development of this scale includes both systematic literature and structural interview, missed out items will be minimized. This will make this scale best outcome measure for documenting patient outcome in India.

ELIGIBILITY:
Inclusion Criteria:

* Preterm and full term neonates with cardio-pulmonary conditions Stable Neonates

Exclusion Criteria:

* Neonates with severe disability Parents who are not wiling to participate their newborn in study

Ages: 28 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates who are suffering from cardio-pulmonary conditions will be taken in the study such as- Respiratory distress syndrome, Pneumonia, Congenital heart defects etc.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Neonatal Cardio-pulmonary outcome measure (N-COM) | Baseline, PRE INTERVENTION, 1 year POST INTERVENTION
  Changes in pre and post Neonatal-cardio-pulmonary outcome measure (N-COM) will be noted. In pulmonary system, cyanosis (peripheral and central cyanosis), nasal grunting, chest retractions, respiratory rate, SPO2, nasal flaring, chest symmetry etc will be checked. In the cardiovascular system, heart rate, pulse rate, congenital heart defects, chest symmetry, heart sounds etc will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Asir J Samuel, MPT, PhD, Study Chair — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Pooja Mehra, BPT, (MPT), Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Neha Sharma, MPT, Study Director — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Maharishi Markandeshwar (M.M) Hospital, Mullana, Ambala, Haryana, Mullana, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided